CLINICAL TRIAL: NCT02294773
Title: Randomized Controlled Trial Evaluating the Timing of Intrauterine Insemination in Relation to the LH Surge
Brief Title: Study Evaluating the Timing of Intrauterine Insemination in Relation to Positive Home Ovulation Prediction Kit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Midwest Fertility Specialists (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: 13-MIDW-101
Record Dates: First submitted 2014-10-01; First posted 2014-11-19 (Estimated); Results first posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-11

CONDITIONS: Infertility
Keywords: Infertility; Intrauterine insemination; Luteinizing hormone surge
MeSH Terms: conditions — Infertility | interventions — Clomiphene; Letrozole

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Day Of (Active Comparator): This group takes either clomiphene or letrozole on cycle days 3-7 and then receives intrauterine insemination on the day the home ovulation predictor kit first turns positive.
  Interventions: Procedure: Intrauterine Insemination; Drug: Clomiphene; Drug: Letrozole
- Day After (Active Comparator): This group takes either clomiphene or letrozole on cycle days 3-7 and then receives intrauterine insemination on the day after the home ovulation predictor kit first turns positive.
  Interventions: Procedure: Intrauterine Insemination; Drug: Clomiphene; Drug: Letrozole

INTERVENTIONS:
Procedure: Intrauterine Insemination — Intrauterine insemination is either performed on the day the home ovulation predictor kit first turns positive or the day after the first positive.
Drug: Clomiphene — Patient is to take clomiphene citrate during cycle days 3-7.
  Other Names: clomid
Drug: Letrozole — Patient is to take letrozole during cycle days 3-7.

SUMMARY:
The aim of this study is to assess the impact of the timing of intrauterine insemination (IUI) in relation to the natural surge of luteinizing hormone (LH), as detected by home ovulation predictor kits, on pregnancy rates per treatment cycle. The study will take place at the offices of Midwest Fertility Specialists and include patients who have been independently recommended by their primary physician to undergo ovulation induction with clomiphene citrate (CC) or letrozole and IUI as therapy for infertility.

DETAILED DESCRIPTION:
Intrauterine insemination is a procedure that is performed in the physician's office. During the procedure the sperm from the male partner are placed directly into the female partner's uterus around the time of ovulation (release of oocyte or egg). Ovulation predictor kits, available over the counter at pharmacies, test for the presence of luteinizing hormone in the urine. When the test result is a positive, it means the hormone is present in the urine. This is a sign of ovulation. Physicians typically choose to perform intrauterine insemination either the day of a positive ovulation test or the day after a positive ovulation test. The purpose of this study is to determine if the day when intrauterine insemination is performed influences the chance of becoming pregnant.

ELIGIBILITY:
Inclusion Criteria:

* All couples consisting of male and female partner undergoing CC or letrozole cycle plus IUI at a single infertility center (Midwest Fertility Specialists)
* The female partner must be aged 21-39
* Infertile couples include those with a diagnosis(s) of unexplained infertility, mild male factor, ovulatory dysfunction, or anovulation
* Evidence of a normal uterus and at least unilateral tubal patency on saline infusion sonogram or hysterosalpingogram within the last 2 years
* Semen analysis for male partner must have minimal sperm concentration of 10 million per milliliter

Exclusion Criteria:

* Recurrent miscarriages
* Nursing mothers
* Diagnoses of primary ovarian failure, diminishing ovarian reserve (as indicated by blood follicle stimulating hormone >10 milliInternationalUnits/mL and/or anti-mullerian hormone level <0.5), abnormal uterine bleeding of undetermined origin, ovarian cyst of undetermined origin, stage IV endometriosis, or sex-hormone dependent tumors
* Documented bilateral tubal obstruction or other uncorrected uterine anomalies (e.g. uterine septum)
* Previous gonadotropin use and/or previous treatment with in vitro fertilization
* Abnormal semen analysis (sperm concentration less than 10 million per mL) or ejaculatory dysfunction in male partner
* Other uncorrected medical condition in female partner that would be a contraindication to attempting elective ovulation induction (e.g., uncontrolled diabetes, intracranial lesion, thyroid or adrenal disease)

Ages: 21 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13 (Actual)
Dates: Start 2013-10; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew Will, MD, Principal Investigator — Midwest Fertility Specialists
Locations (2):
- United States (2):
  - Midwest Fertility Specialists- Fort Wayne, Fort Wayne, Indiana
  - Midwest Fertility Specialists, Indianapolis, Indiana

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Patients recruited from two clinical offices from 1/2014 until 9/2015.
Groups:
- Insemination Day Of Positive OPK: This group takes either clomiphene or letrozole on cycle days 3-7 and then receives intrauterine insemination on the day the home ovulation predictor kit first turns positive.
  Intrauterine Insemination: Intrauterine insemination is either performed on the day the home ovulation predictor kit first turns positive or the day after the first positive.
  Clomiphene: Patient is to take clomiphene citrate during cycle days 3-7.
  Letrozole: Patient is to take letrozole during cycle days 3-7.
- Insemination Day After Positive OPK: This group takes either clomiphene or letrozole on cycle days 3-7 and then receives intrauterine insemination on the day after the home ovulation predictor kit first turns positive.
  Intrauterine Insemination: Intrauterine insemination is either performed on the day the home ovulation predictor kit first turns positive or the day after the first positive.
  Clomiphene: Patient is to take clomiphene citrate during cycle days 3-7.
  Letrozole: Patient is to take letrozole during cycle days 3-7.
Period: Overall Study
Arm/Group | Insemination Day Of Positive OPK | Insemination Day After Positive OPK
Started | 7 | 6
Completed | 7 | 4
Not Completed | 0 | 2
Not completed — Withdrawal by Subject | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Insemination Day Of Positive OPK | Insemination Day After Positive OPK | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.4 (5.9) | 29.6 (3.05) | 30.1 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7 | 6 | 13
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13
Body Mass Index [Mean (Standard Deviation); unit: kg/m^2] | 30 (8.9) | 25 (4) | 27.9 (7.5)
Day 3 Follicle Stimulating Hormone [Mean (Standard Deviation); unit: mIU/ml] | 7.6 (1.7) | 6.2 (1.9) | 6.9 (1.8)
Anti-mullerian Hormone [Mean (Standard Deviation); unit: ng/ml] | 3.1 (2.2) | 5.8 (0) | 5.2 (2.3)
Sperm Concentration [Mean (Standard Deviation); unit: million sperm/ml] | 32.6 (13.9) | 71.2 (39.2) | 39.4 (30.9)
Sperm morphology [Mean (Standard Deviation); unit: Percent normal] | 5.6 (2.3) | 8.5 (2.4) | 6.2 (2.6)
Mid-luteal progesterone [Mean (Standard Deviation); unit: ng/ml] | 21.1 (16.4) | 12.1 (4.3) | 18.6 (13.7)

OUTCOME MEASURES:

1. Primary Outcome: Number of Pregnancies Achieved Per Menstrual Cycle.
Time Frame: Up to 3 months
Measure: Number; unit: pregnancies per cycle
Arm/Group | Insemination Day Of Positive OPK | Insemination Day After Positive OPK
Number analyzed (Participants) | 7 | 6
pregnancies per cycle | 0 | 0

2. Other Pre Specified Outcome: Per Cycle Pregnancy Rate Based on Infertility Diagnosis
Time Frame: Up to cycle day 35
Measure: Number; unit: pregnancies per cycle
Arm/Group | Insemination Day Of Positive OPK | Insemination Day After Positive OPK
Number analyzed (Participants) | 7 | 6
pregnancies per cycle | 0 | 0

3. Other Pre Specified Outcome: Pregnancy Rate Per Female Partner Age
Description: Pregnancy rate will be compared between patients <35 and >35 at time of study entry.
Time Frame: Up to cycle day 35
Measure: Number; unit: pregnancies per cycle
Arm/Group | Insemination Day Of Positive OPK | Insemination Day After Positive OPK
Number analyzed (Participants) | 7 | 6
pregnancies per cycle
  Female age < 35 | 0 | 0
  Female age > 35 | 0 | 0

4. Other Pre Specified Outcome: Pregnancy Rate Per Semen Morphology Score
Description: Comparison of pregnancy rate based on semen morphology of <4% vs >4% normal morphology scores.
Time Frame: Up to cycle day 35
Measure: Number; unit: pregnancies per cycle
Arm/Group | Insemination Day Of Positive OPK | Insemination Day After Positive OPK
Number analyzed (Participants) | 7 | 6
pregnancies per cycle
  Semen morphology < 4% | 0 | 0
  Semen morphology > 4% | 0 | 0

5. Other Pre Specified Outcome: Pregnancy Rate Per Body Mass Index Category
Time Frame: Up to cycle day 35
Measure: Number; unit: pregnancies per cycle
Arm/Group | Insemination Day Of Positive OPK | Insemination Day After Positive OPK
Number analyzed (Participants) | 7 | 6
pregnancies per cycle
  Body mass index normal | 0 | 0
  Body mass index overweight | 0 | 0
  Body mass index obese | 0 | 0

ADVERSE EVENTS:
Arm/Group | Insemination Day Of Positive OPK | Insemination Day After Positive OPK
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 0/6

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes